CLINICAL TRIAL: NCT00790322
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Phase III Clinical Study to Assess the Efficacy and Safety of SBG on Oral Mucositis in Head and Neck Cancer Patients Undergoing Radiation Therapy With or Without Chemotherapy
Brief Title: Efficacy and Safety Study of SBG vs Placebo in Head and Neck Cancer Patients Undergoing Radiation Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biotec Pharmacon ASA (Industry)
Responsible Party: Vice President Clinical Development, Biotec Pharmacon ASA
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SBG-2-03; EudraCT-number: 2008-002340-42
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2010-02

CONDITIONS: Head and Neck Cancer; Oral Mucositis
Keywords: Cancer; Radiation therapy; Radiotherapy; Oral Mucositis; SBG
MeSH Terms: conditions — Head and Neck Neoplasms; Stomatitis; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental)
  Interventions: Drug: SBG
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SBG — Soluble beta-1,3/1,6-glucan is a solution for oral use
  Arms: Active
Other: Placebo — Solution for oral use
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of SBG vs placebo on oral mucositis in head and neck cancer patients undergoing radiation therapy.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the efficacy and safety of soluble beta-1,3/1,6-glucan (SBG) on oral mucositis compared to placebo in head and neck cancer patients undergoing radiation therapy with or without chemotherapy.

ELIGIBILITY:
* Patients with a normal oral mucosa who is scheduled to receive radiation therapy for their head and neck cancer will be enrolled into the study.
* Patients with previous head and neck cancer and/or radiation therapy in the head and neck area and history/clinical evidence of active significant acute or chronic conditions that may compromise the ability to evaluate or interpret the effects of the study treatment on mucositis will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2008-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Compare the proportion of patients in the two arms who develop severe oral mucositis | During radiation therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Institute Gustave Roussy, Villejuif Cédex, France